CLINICAL TRIAL: NCT00913991
Title: Mechanisms of the Relaxation Response in Elderly Hypertensives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Dusek, Jeffery, Research Director, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R21AT003315-01 (NIH)
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2010-02

CONDITIONS: Hypertension
Keywords: Nitric Oxide
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stress Management #1 (Experimental): 8 weeks of individual stress management training sessions
  Interventions: Behavioral: Stress Management Training
- Stress Management #2 (Active Comparator): 8 weeks of individual stress management training sessions
  Interventions: Behavioral: Stress Management Training

INTERVENTIONS:
Behavioral: Stress Management Training — Weekly 60-minute session with a trainer for 8 consecutive weeks. Daily home practice of approximately 20 minutes per day via CD.
  Arms: Stress Management #1
Behavioral: Stress Management Training — Weekly 60-minute session with a trainer for 8 consecutive weeks. Daily home practice of approximately 20 minutes per day via CD.
  Arms: Stress Management #2

SUMMARY:
Systolic Hypertension is a disorder which is characterized by significant elevations in systolic blood pressure in association with normal diastolic blood pressure. Typically, this develops in individuals >50 years of age and is associated with an increased risk of stroke and myocardial infarction. While there are many effective therapies for essential/diastolic hypertension, the treatment of systolic hypertension is complicated by side effects from traditional therapies. This limits therapeutic options and has resulted in a number of at-risk individuals being left untreated.

We are conducting a randomized, controlled trial (n=90) to compare the effects of two different stress management training on blood pressure. The primary outcome is change in systolic blood pressure and pulse pressure. Secondary outcomes are changes in nitric oxide, stress hormones and psychological well-being. Additional analyses will be conducted to assess for other confounding effects on BP and PP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; stage I SH (140-159 mm Hg SBP and < 90 mm Hg DBP), > 55 years of age; taking at least 1 anti-hypertensive medication at a stable dose for 1 month preceding the screening visit; understanding of English; normal hearing; and able to provide informed consent.

Exclusion Criteria:

* Presence of current neurological, psychiatric, medical or musculoskeletal disorder; current asthma; severe seasonal allergies resulting in screening NO values > 60 ppb; current smoking; experience with yoga, meditation, guided imagery or other techniques that evoke the RR; hematocrit below 32; glucose lower than 50 or higher than 200; a creatinine greater than 1.3, Mini-Mental Status Exam score less than 26 or clinical depression based on a score of greater than 15 on the CES-D and Health Counselor's clinical evaluation. Subjects can not take the following medications: beta-agonist bronchodilators, systemic corticosteroids, anti-convulsants, immunosuppressive or cytotoxic therapy (currently or within the last 12 months), anabolic steroids, anti-depressants (not including SSRIs), anti-psychotics, chronic sypathomimetic medications, and dicyclomine.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 8 weeks

SECONDARY OUTCOMES:
Nitric Oxide and epinephrine levels | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Dusek, PhD, Principal Investigator — Allina Health System
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States